CLINICAL TRIAL: NCT04539938
Title: A Single Arm, Open Label Phase 2 Study of Tucatinib in Combination With Trastuzumab Deruxtecan in Subjects With Previously Treated Unresectable Locally-Advanced or Metastatic HER2+ Breast Cancer
Brief Title: A Study of Tucatinib Plus Trastuzumab Deruxtecan in HER2+ Breast Cancer
Acronym: HER2CLIMB-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGNTUC-025; C4251006 (Other: Alias Study Number)
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: HER2 Positive Breast Cancer
Keywords: HER2+ breast cancer; Metastatic breast cancer; Stage IV breast cancer; Seattle Genetics
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Tucatinib + trastuzumab deruxtecan
  Interventions: Drug: tucatinib; Drug: trastuzumab deruxtecan

INTERVENTIONS:
Drug: tucatinib — 300 mg orally twice daily
  Other Names: TUKYSA, ARRY-380, ONT-380; PF-07265792
Drug: trastuzumab deruxtecan — 5.4 mg/kg via intravenous (into the vein; IV) infusion on Day 1 of each of 21-day cycle
  Other Names: T-DXd, Enhertu, DS-8201

SUMMARY:
This trial studies how well the drug tucatinib works when given with trastuzumab deruxtecan (T-DXd). It will also look at what side effects happen when these drugs are given together. A side effect is anything a drug does besides treating cancer.

Participants in this trial have HER2-positive (HER2+) breast cancer that has either spread to other parts of the body (metastatic) or cannot be removed completely with surgery (unresectable). All participants will get both tucatinib and T-DXd.

ELIGIBILITY:
Inclusion Criteria

* Have confirmed HER2+ breast cancer, as defined by the current American Society of Clinical Oncology - College of American Pathologists (ASCO/CAP) guidelines, previously determined at a Clinical Laboratory Improvements Amendments (CLIA)-certified or International Organization for Standardization (ISO)-accredited laboratory.
* History of prior treatment with a taxane and trastuzumab in the LA/M setting OR progressed within 6 months after neoadjuvant or adjuvant treatment, including a taxane and trastuzumab.
* Have progression of unresectable LA/M breast cancer after last systemic therapy (as confirmed by investigator), or be intolerant of last systemic therapy
* Have measurable disease assessable by RECIST v1.1
* Have Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1
* Have a life expectancy of at least 6 months, in the opinion of the investigator
* CNS Inclusion - Based on medical history and screening contrast brain magnetic resonance imaging (MRI), participants with a history of brain metastases must have one of the following:

  * Untreated brain metastases not needing immediate local therapy. For participants with untreated central nervous system (CNS) lesions >2.0 cm on screening contrast brain MRI, discussion with and approval from the medical monitor is required prior to enrollment
  * Previously treated brain metastases

    * Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local CNS therapy, provided that there is no clinical indication for immediate re-treatment with local therapy in the opinion of the investigator
    * Participants treated with CNS local therapy for newly identified or previously treated progressing lesions found on contrast brain MRI performed during screening for this study may be eligible to enroll if all of the following criteria are met:

      * Time since whole brain radiation therapy (WBRT) is ≥14 days prior to first dose of study treatment, time since stereotactic radiosurgery (SRS) is ≥7 days prior to first dose of study treatment, or time since surgical resection is ≥28 days
      * Other sites of measurable disease by RECIST v1.1 are present
    * Relevant records of any CNS treatment must be available

Exclusion Criteria

* Have previously been treated with:

  * Lapatinib or neratinib within 12 months of starting study treatment (except in cases where lapatinib or neratinib was given for ≤21 days and was discontinued for reasons other than disease progression or severe toxicity)
  * Tucatinib or enrolled on a tucatinib clinical trial
  * Any investigational HER2/epidermal growth factor receptor (EGFR) or HER2 tyrosine kinase inhibitor (TKI) (eg, afatinib) at any time previously
  * Trastuzumab deruxtecan or another antibody-drug conjugate (ADC) consisting of an exatecan derivative
* Have received treatment with:

  * Any systemic anti-cancer therapy (including hormonal therapy) or experimental agent ≤21 days of first dose of study treatment or are currently participating in another interventional clinical trial. An exception for the washout of hormonal therapies is gonadotropin releasing hormone (GnRH) agonists used for ovarian suppression in premenopausal women, which are permitted concomitant medications
  * Treatment with non-CNS radiation ≤7 days prior to first dose of study treatment
  * Major surgery <28 days of first dose of study treatment
* Have clinically significant cardiopulmonary disease (such as history of iterstitial lung disease (ILD)/pneumonitis that required systemic corticosteroids, or have current ILD/pneumonitis, or where suspected ILD /pneumonitis cannot be ruled out be imaging at screening)
* Have known myocardial infarction or unstable angina within 6 months prior to first dose of study treatment
* Known to be positive for hepatitis B by surface antigen expression. Known to be positive for hepatitis C infection. Participants who have been treated for hepatitis C infection are permitted if they have documented sustained virologic response of 12 weeks
* Presence of known chronic liver disease
* Active or uncontrolled clinically serious infection
* Have inability to swallow pills or significant gastrointestinal disease which would preclude the adequate oral absorption of medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (132):
- United States (132):
  - University Of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, IDS Pharmacy, Birmingham, Alabama
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - UCLA Hematology/Oncology - Alhambra, Alhambra, California
  - UCLA Hematology/Oncology - Burbank, Burbank, California
  - City of Hope (City of Hope National Medical Center, City of Hope Medical center), Duarte, California
  - City of Hope Investigational Drug Services (IDS), Duarte, California
  - UCLA Hematology/Oncology - Laguna Hills, Laguna Hills, California
  - (IRB# 20-001502) Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/Oncology - Pasadena, Pasadena, California
  - Zuckerberg San Francisco General Hospital- Breast Clinic, San Francisco, California
  - Zuckerberg San Francisco General Hospital- Oncology Clinic, San Francisco, California
  - University of California, San Francisco (UCSF) Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCLA Hematology/Oncology - San Luis Obispo, San Luis Obispo, California
  - UCLA Hematology/Oncology - Santa Barbara, Santa Barbara, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - UCLA Hematology/Oncology Parkside, Santa Monica, California
  - UCLA Hematology/Oncology - Ventura, Ventura, California
  - UCLA Hematology/Oncology - Westlake, Westlake Village, California
  - University of Colorado Denver CTO/CTRC - Outpatient., Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - UC Health Lone Tree Medical Center, Lone Tree, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Lecanto, Florida
  - Florida Cancer Specialists, Ocala, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, The Villages, Florida
  - Florida Cancer Specialists, Trinity, Florida
  - Florida Cancer Specialists, Winter Park, Florida
  - Northside Hospital, Inc - GCS/Athens, Athens, Georgia
  - Winship Cancer Institute @ Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Cancer Care - Atlanta, Atlanta, Georgia
  - Northside Hospital, Inc. - Central Research Department, Atlanta, Georgia
  - Northside Hospital, Inc. - GCS/Center Pointe, Atlanta, Georgia
  - Northside Hospital, Inc - GCS/Blairsville, Blairsville, Georgia
  - Northside Hospital, Inc - GCS/Canton, Canton, Georgia
  - Atlanta Cancer Care - Cumming, Cumming, Georgia
  - Northside Hospital, Inc. - GCS/Decatur, Decatur, Georgia
  - NHCI Suburban Hematology-oncology Associates - Duluth, Duluth, Georgia
  - NHCI Suburban Hematology-oncology Associates - lawrenceville, Lawrenceville, Georgia
  - Northside Hospital, Inc - GCS/Macon, Macon, Georgia
  - Northside Hospital, Inc. - GCS/Marietta, Marietta, Georgia
  - Atlanta Cancer Care - Stockbridge, Stockbridge, Georgia
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute- Chestnut Hill, Newton, Massachusetts
  - Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, PA, Coon Rapids, Minnesota
  - Mercy Hospital - Unity Campus, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Allina Health Cancer institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Allina Health Cancer Institute, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA, Saint Paul, Minnesota
  - Minnesota Oncology Hematology, PA, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Papillion, Nebraska
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - Investigational Drug Service Pharmacy, Long Island City, New York
  - Evelyn H. Lauder Breast and Imaging Center (BAIC)., New York, New York
  - MSK Nassau, Uniondale, New York
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - UPMC Hillman Cancer Center Passavant North, Cranberry Township, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Hillman Cancer Center Mountainview, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center UPMC East, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center Upper Saint Clair, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute Investigational Drug Service UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers William M. Cooper Ambulatory Care Pavilion of the Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center UPMC Passavant, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center Uniontown, Uniontown, Pennsylvania
  - UPMC Hillman Cancer Center Washington, Washington, Pennsylvania
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Cleveland, Tennessee
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hendersonville, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - U.T. MD Anderson Cancer Center, Houston, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology lnvestigational Products Center (IPC), Irving, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Virginia Cancer Specialists, PC, Leesburg, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Low Moor, Virginia
  - Virginia Cancer Specialists, PC, Reston, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Salem, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc. D.B.A Blue Ridge Cancer Care, Wytheville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - UW Health Oncology - One South Park, Madison, Wisconsin
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNTUC-025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with unresectable locally advanced or metastatic (LA/M) human epidermal growth factor receptor 2 positive (HER2+) breast cancer with or without brain metastases, who received prior treatment with a taxane and trastuzumab or progressed within 6 months after neoadjuvant or adjuvant treatment involving a regimen including a taxane and trastuzumab (with or without pertuzumab) were enrolled at 24 sites in the United States.
Pre-assignment Details: A total of 94 participants were screened of which 24 failed screening and 70 participants were enrolled in the study. Results are presented for primary outcome measures at data cutoff 15 July 2024 (primary completion date [PCD]). Remaining outcome measures would be reported upon completion of their analyses at study completion date.
Groups:
- Total Participants: Participants with HER2+ LA/mBC with or without history of brain metastases received tucatinib 300 milligram (mg) orally (PO) twice daily (BID) on Days 1 to 21 and Trastuzumab Deruxtecan (T-DXd) 5.4 milligram per kilogram (mg/kg) intravenous (IV) on Day 1 of each 21-day cycle. Participants received treatment until unacceptable toxicity, progressive disease (PD), investigator or participants decision to discontinue, or study closure.
Period: Overall Study
Arm/Group | Total Participants
Started | 70
Completed | 36
Not Completed | 34
Not completed — Death | 30
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: The all-treated participants analysis set included all participants who receive any amount of study drug (tucatinib and/or trastuzumab deruxtecan).
Groups:
- Total Participants: Participants with HER2+ LA/mBC with or without history of brain metastases received tucatinib 300mg PO BID on Days 1 to 21 and Trastuzumab Deruxtecan (T-DXd) 5.4 mg/kg IV on Day 1 of each 21-day cycle. Participants received treatment until unacceptable toxicity, PD, investigator or participants decision to discontinue, or study closure.
Arm/Group | Total Participants
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 56
  More than one race | 0
  Unknown or Not Reported | 2
Presence or history of treated or untreated brain metastases [Count of Participants; unit: Participants]
  Yes | 27
  No | 43
HER2 testing results [Count of Participants; unit: Participants]
  Immunohistochemistry (IHC) 3 plus (+) | 41
  IHC 2+ and/or Fluorescence in situ hybridization + | 28
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (cORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 According to Investigator (INV) Assessment
Description: Confirmed objective response rate was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) per investigator according to RECIST v1.1. For a response to be considered confirmed, the subsequent response had to be at least 4 weeks after the initial response. CR: disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). PR: a greater than equal to (>=) 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. 95% exact confidence interval (CI) was based on Clopper-Pearson method.
Time Frame: From the first dose of study treatment until the first documented PD or before start of any new anti-cancer therapy (up to 43 months)
Population: Response-evaluable analysis set included all participants with measurable disease who (1) had a baseline disease assessment, (2) received at least one dose of study drug (tucatinib and/or trastuzumab deruxtecan), and (3) had at least 1 post-baseline assessment or discontinued treatment due to PD, clinical progression, toxicity, or death.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Total Participants
Number analyzed (Participants) | 70
Percentage of participants | 51.4 [39.2 to 63.6]

2. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1 According to INV
Description: PFS as per INV was defined as the time from the start of the study treatment to the first documentation of PD per RECIST v1.1 or death due to any cause, whichever occurred first. PD: at least a 20 % increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From the start of study treatment until the first documentation of PD or death, whichever occurred first
Population: The all treated participants includes all participants who received any amount of study drug (tucatinib and/or trastuzumab deruxtecan).
Reporting Status: Not Posted, anticipated posting 2026-12

3. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 According to INV
Description: DOR was defined the time from the date of the first documented objective response (CR or PR that is subsequently confirmed) to the date of the first documented PD per RECIST v1.1 or death due to any cause, whichever occurred first. PD: at least a 20 % increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. CR: disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: a >= 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From the first documented objective response until the first documentation of PD or death, whichever occurred first
Population: The response-evaluable analysis set included all participants with measurable disease who (1) had a baseline disease assessment, (2) received at least one dose of study drug (tucatinib and/or trastuzumab deruxtecan), and (3) had at least 1 post-baseline assessment or discontinued treatment due to PD, clinical progression, toxicity, or death.
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1
Description: DCR was defined as the percentage of participants with confirmed CR, PR or stable disease (SD) or non-CR/non-PD per RECIST v1.1. CR: disappearance of all target lesions and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: a >= 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From the first dose study treatment until PD or death, whichever occurred first
Population: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of study treatment to the date of death due to any cause.
Time Frame: From date of start of study treatment until date of death or censoring date
Population: The all-treated participants included all participants who received any amount of study drug (tucatinib and/or trastuzumab deruxtecan).
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib or trastuzumab deruxtecan) and up through 30 days after the last dose of study treatment.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment
Population: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was an AE that at any dose, met any of the following criteria: resulted in death, was life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or disability (substantial disruption of the participant's ability to conduct normal life functions), congenital anomaly/birth defect or considered medically significant.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: Number of Participants With Adverse Events Based on Severity
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib or trastuzumab deruxtecan) and up through 30 days after the last dose of study treatment. AEs were graded based on National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0 criteria where, grade 1= mild; grade 2= moderate; grade 3= severe; grade 4= life-threatening; grade 5= death.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: Number of Participants With Treatment Related Adverse Events
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. Relatedness of AEs to study treatment was determined by the investigator.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2026-12

10. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Following laboratory parameters will be assessed: Serum chemistry included: bicarbonate, blood urea nitrogen, calcium, creatinine, chloride, glucose, magnesium, phosphorus, potassium, and sodium. liver function tests (LFTs) include albumin, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (and both direct and indirect bilirubin when total bilirubin is > upper limit of normal (ULN), and total protein. white blood cell counts with 5-part differential (neutrophils, lymphocytes, monocytes, eosinophils, and basophils), platelet count, hemoglobin, and hematocrit. Coagulation: international normalized ratio (INR), prothrombin time (PT), and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT), A serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment
Population: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-12

11. Secondary Outcome: Number of Participants With TEAEs Leading to Dose Modification
Description: An AE was defined was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. A TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib or trastuzumab deruxtecan) and up through 30 days after the last dose of study treatment. Participants experienced tucatinib dose modification due to TEAEs. Dose modification included dose reduction, dose delay, dose hold, drug interruption.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment
Population: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-12

12. Secondary Outcome: Number of Participants With TEAEs Leading to Treatment Discontinuation
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment
Population: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-12

13. Secondary Outcome: Change From Baseline in Ejection Fraction
Description: Cardiac ejection fraction will be assessed using multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
Time Frame: Baseline and end of treatment
Population: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-12

14. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital signs will include body temperature, respiratory rate, heart rate, and systolic and diastolic blood pressure.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment
Population: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: From start of study treatment (Day 1) up to 30 days after last dose of study treatment (approximately up to 43.5 months)
Description: Same event may appear as both non-serious adverse event and serious adverse event (SAE); however, are presented as distinct events. Event may be categorized as serious in 1 participant and non-serious in another or may have experienced both SAE and non-SAE. The all-treated participants analysis set included all participants who received any amount of study drug (tucatinib and/or trastuzumab deruxtecan).
Arm/Group | Total Participants
All-Cause Mortality (participants affected / at risk) | 33/70
Serious Adverse Events (participants affected / at risk) | 25/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Participants (N=70)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Tooth infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Participants (N=70)
Anaemia (Blood and lymphatic system disorders) | 7 (8)
Neutropenia (Blood and lymphatic system disorders) | 5 (14)
Dry eye (Eye disorders) | 5 (6)
Vision blurred (Eye disorders) | 11 (12)
Abdominal pain (Gastrointestinal disorders) | 9 (16)
Constipation (Gastrointestinal disorders) | 37 (59)
Diarrhoea (Gastrointestinal disorders) | 55 (103)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8)
Haemorrhoids (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 54 (90)
Stomatitis (Gastrointestinal disorders) | 10 (12)
Vomiting (Gastrointestinal disorders) | 42 (68)
Chills (General disorders) | 7 (7)
Fatigue (General disorders) | 50 (64)
Influenza like illness (General disorders) | 5 (6)
Malaise (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 8 (10)
Pyrexia (General disorders) | 7 (9)
COVID-19 (Infections and infestations) | 11 (11)
Conjunctivitis (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 11 (14)
Urinary tract infection (Infections and infestations) | 17 (34)
Fall (Injury, poisoning and procedural complications) | 7 (7)
Alanine aminotransferase increased (Investigations) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 6 (8)
Blood bilirubin increased (Investigations) | 4 (11)
Blood creatinine increased (Investigations) | 5 (8)
Neutrophil count decreased (Investigations) | 8 (11)
Weight decreased (Investigations) | 15 (16)
Weight increased (Investigations) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 25 (32)
Dehydration (Metabolism and nutrition disorders) | 8 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (29)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Dizziness (Nervous system disorders) | 10 (14)
Dysgeusia (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 21 (32)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (11)
Insomnia (Psychiatric disorders) | 8 (8)
Dysuria (Renal and urinary disorders) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (17)
Rash (Skin and subcutaneous tissue disorders) | 5 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Hot flush (Vascular disorders) | 8 (9)
Hypotension (Vascular disorders) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04539938/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT04539938/SAP_001.pdf